CLINICAL TRIAL: NCT01924091
Title: Comparison of the Pharmacokinetics and Pharmacodynamics of Single Dose Dapivirine Vaginal Gel and Film Formulation
Brief Title: PK/PD of Single Dose Dapivirine Vaginal Film
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FAME-02B; DAIDS-ES# 11939 (Other: DAIDS)
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Pharmaokinetics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapivirine Gel (Experimental): As outlined above, multiple gel formulations of dapivirine have been developed for vaginal use.
  Three formulations, Dapivirine Gel-001 (Gel-001), Dapivirine Gel-002 (Gel-002), and Dapivirine Gel 4750 (Gel 4750) are no longer in development. Dapivirine Gel 4789, which has been tested in one clinical trial (IPM012), and Dapivirine Gel 4759 were recently evaluated in clinical trials, IPM 014A and IPM 020. This trial will use Dapivirine Gel 4759.
  Interventions: Drug: Dapivirine gel
- Dapivirine Film (Experimental): Dapivirine film is formulated in a polyvinyl alcohol (PVA) based vaginal film containing hydroxypropyl methyl cellulose (HPMC) E5 (5 cp), polyethylene glycol 8000 (PEG), propylene glycol, and glycerin. PVA constituted 55.1% (w/w) of the film. The target loading dose for the film is 1.25 mg dapivirine per film based on phase I studies using dapivirine gels at concentrations of 0.01%, 0.02% and 0.05%30-33. The quantity of gel administered in these studies was 2.5 mL. Consequently the administered dose corresponds to 0.25, 0.5 and 1.25 mg dapivirine, respectively.
  Interventions: Drug: Dapivirine film

INTERVENTIONS:
Drug: Dapivirine gel
  Arms: Dapivirine Gel
Drug: Dapivirine film
  Arms: Dapivirine Film

SUMMARY:
To compare drug concentrations in vaginal fluid, genital tissue, and blood

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older with a history of receptive vaginal intercourse.
2. HIV negative by EIA within 28 days of enrollment.
3. Understand and agree to local STI reporting requirements.
4. Able and willing to provide written informed consent to take part in the study.
5. Able and willing to provide adequate information for locator purposes.
6. Availability to return for all study visits, barring unforeseen circumstances.
7. Availability to return for the second formulation dosing at the same time in the subject's menstrual cycle as when the first formulation was administered, at least 10 days before menses.
8. Willing to abstain from vaginal intercourse and insertion of anything (e.g., drug, vaginal douche, or sex toy) in vagina for 72 hours before each study product exposure, and 7 days following each vaginal sampling procedure.
9. Willingness to have partner(s) use condoms (must not contain Nonoxynol-9) for the duration of the study.
10. Agree not to participate in other research studies involving drugs and/or medical devices.
11. Negative qualitative urine pregnancy test.
12. Per participant report, using an effective method of contraception at enrollment; hormonal method (except vaginal ring) used continuously for the past 30 days; intrauterine device (IUD [copper or hormonal] inserted at least 30 days prior to enrollment); female sterilization; abstinent from sexual activity with male partner for the past 30 days; or sexual activity with vasectomized partner; and willingness to use effective method of contraception until the completion of final scheduled study visit if enrolled.
13. Willingness to remain in the research unit for up to 24 hours on each of two dosing days, -

Exclusion Criteria:

1. Current sexual partner known by participant to be HIV seropositive.
2. Individuals who, by history, engage in condom-less intercourse with HIV-infected partners, or partners that have unknown HIV serostatus, or women who exchange sex for money, shelter, or gifts.
3. Active sexually transmitted infection or documented treatment of sexually transmitted infections including, but not limited to: chlamydia, gonorrhea, syphilis, trichomonas, cervicitis or PID within 6 months prior to enrollment.
4. Known history of genital HSV (diagnosed by either clinical or laboratory test).
5. Symptomatic vaginal candidiasis or bacterial vaginosis.
6. Undiagnosed irregular uterine bleeding
7. Pathology of the female genital tract, which in the judgment of the investigator might increase the risk of the study to the research participant.
8. Individuals who are status post hysterectomy.
9. History of any cervicovaginal procedure (i.e. colposcopy with cervical biopsy) within the past 2 months. Individuals who have a history of cone biopsy or extensive loop electrosurgical excision procedure (LEEP), which in the judgment of the investigator may affect permeability assessment.
10. Any known primary or secondary uro-genital malformations, which in the assessment of the investigator may interfere with the intended urine collection for PK studies.
11. Use of vaginally administered medications within 4 week of enrollment
12. Any active urinary tract infection
13. By history, subjects with irregular menstrual cycles.
14. At screening:

    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 1.5 X the site laboratory ULN (upper limit of normal)
    * Hemoglobin less than 10.0 g/dL
    * Platelet count less than 100,000/mm3
    * Other safety tests outside of the normal range that in the judgment of the investigator may interfere with conduct of the study.
    * Positive findings on urinalysis that are clinically significant in the opinion of the investigator
15. Estimated creatinine clearance < 60 ml/min based on established nomograms
16. Recent history (past 6 months) of injection drug use or, a level of alcohol use that, in the judgement of the Investigator of Record, may interfere with the conduct of this study.
17. Unwillingness to refrain from aspirin and NSAIDs product use for one week prior to and one week post study procedures.
18. Use of warfarin or heparin.
19. Use of systemic immunomodulatory medications within 4 weeks of enrollment.
20. Use of product containing nonoxynol-9 within 4 weeks of enrollment.
21. Use of any investigational products within 4 weeks of enrollment.
22. Any other medical conditions deemed not safe for participation by the investigator.
23. Any individual that is actively breast feeding.
24. Post-menopausal defined as 12 months of amenorrhea.

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Dapivirine concentrations in plasma | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Principal Investigator — John's Hopkins University